CLINICAL TRIAL: NCT03303482
Title: A Randomized Controlled Trial of Trauma-awareness Training for Early Childhood Educators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: United Way of Greater Philadelphia and Southern New Jersey (UWGPSNJ) (Unknown); Lakeside Global Institute (Other); The School District of Philadelphia (Other)
Responsible Party: Principal Investigator, Robert Whitaker, Professor of Epidemiology and Biostatistics and Pediatrics, Temple University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UW17246
Record Dates: First submitted 2017-09-18; First posted 2017-10-06 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Burnout, Professional
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Intervention Model Description: The investigators will randomly assign consenting teachers by classroom (lead teacher and/or assistant teacher) to either the fall or spring course (intervention and waitlist control groups, respectively). The course will be taught to groups of 16 teachers, with four groups in the fall course (64 teachers) and four in the spring course (64 teachers). To determine the impacts of the training intervention on those assigned to the fall course (intervention groups), those assigned to the spring course (control groups) will serve as concurrent controls during the fall.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Behavioral: Enhancing Trauma Awareness (Diane Wagenhals, MEd-Lakeside Global Institute)
- Waitlist Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Enhancing Trauma Awareness (Diane Wagenhals, MEd-Lakeside Global Institute) — The trauma awareness professional development course is delivered in a small group (up to 16 participants; 2.5 hours every other week over 12 weeks). The course provides an environment for professionals to explore in depth the complex nature of trauma, while also recognizing and emphasizing the highly sensitive nature of trauma that is essential to becoming trauma-informed. The course facilitates a heightened awareness and appreciation for trauma-related behaviors and consequences that influence relationships and systems and that persist across generations.
  Arms: Intervention Group

SUMMARY:
Background. To increase school readiness, Pre-K programs for low-income children must be responsive to the role of trauma in the lives of children, families, and staff. In 2017-2018, the School District of Philadelphia's (SDP) Office of Early Childhood Education will help Pre-K teachers support children's social-emotional and behavioral health, which is essential for early learning, by offering teachers a professional development course called Enhancing Trauma Awareness (ETA).

Purpose. To determine whether teachers who take ETA will have: 1) better work functioning; 2) more trusting work relationships; and 3) better health.

Population. Pre-K classroom teachers (n=128) working in centers under SDP auspice that serve exclusively low-income (≤300 % of poverty) children.

Intervention. A 12-week professional development course-Enhancing Trauma Awareness-will delivered by Lakeside Global Institute in 6 group sessions, with 16 teachers per group and each session lasting 2.5 hours.

Design. Consenting teachers will be randomly assigned by classroom (lead teacher and/or assistant teacher) to receive the ETA course in either fall 2017 (intervention groups) or spring 2018 (wait-list control groups).

Data collection and analysis. An external evaluation team (Temple University) will administer a confidential, online survey to all 128 teachers in fall 2017 (before fall course), winter 2017 (after fall course), and spring 2018 (after spring course). Teacher-children relationship quality will be the a priori primary outcome, and secondary outcomes will be assessed across the domains of work functioning, trust, and health.

ELIGIBILITY:
Inclusion Criteria:Preschool classroom teacher who works in a center that is under the auspice of the School District of Philadelphia and serves exclusively low-income (≤300 % of poverty) children.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Change in teacher-children relationship quality (specifically, levels of perceived conflict) at 3 months | The teacher-children relationship quality measurement will be assessed for all 128 teachers through online surveys at baseline (before the fall course) and at 3 months (after the fall course).
  A modified version of the Student-Teacher Relationship Scale (STRS) conflict subscale will be used to allow each teacher to provide one global or aggregated assessment of her/his relationships with all the children in the classroom. The conflict subscale includes eight items to assess negative, insecure, and hostile aspects of relationships.

SECONDARY OUTCOMES:
Change in mindfulness (Cognitive and Affective Mindfulness Scale-Revised) at 3 months | The measure will be assessed for all 128 teachers through online surveys at baseline (before the fall course) and at 3 months (after the fall course).
Change in empathy (Interpersonal Reactivity Index) at 3 months | The measure will be assessed for all 128 teachers through online surveys at baseline (before the fall course) and at 3 months (after the fall course).
Change in emotion regulation (Emotion Regulation Questionnaire) at 3 months | The measure will be assessed for all 128 teachers through online surveys at baseline (before the fall course) and at 3 months (after the fall course).
Change in compassion satisfaction (Professional Quality of Life Scale) at 3 months | The measure will be assessed for all 128 teachers through online surveys at baseline (before the fall course) and at 3 months (after the fall course).
Change in job satisfaction (adapted from Gallup Well-Being Work Index) at 3 months | The measure will be assessed for all 128 teachers through online surveys at baseline (before the fall course) and at 3 months (after the fall course).
Change in attitudes about trauma-informed care (Attitudes Related to Trauma-Informed Care Scale) at 3 months | The measure will be assessed for all 128 teachers through online surveys at baseline (before the fall course) and at 3 months (after the fall course).
Change in burnout (Maslach Burnout Inventory General) at 3 months | The measure will be assessed for all 128 teachers through online surveys at baseline (before the fall course) and at 3 months (after the fall course).
Change in trust in relationships with parents, supervisors, and other staff members (adapted from Trust in Schools Instruments) at 3 months | The measure will be assessed for all 128 teachers through online surveys at baseline (before the fall course) and at 3 months (after the fall course).
Change in mentally and physically unhealthy days (CDC Health-Related Quality of Life Healthy Days Core Module) at 3 months | The measure will be assessed for all 128 teachers through online surveys at baseline (before the fall course) and at 3 months (after the fall course).
Change in quality and duration of nighttime sleep (Pittsburgh Sleep Quality Index) at 3 months | The measure will be assessed for all 128 teachers through online surveys at baseline (before the fall course) and at 3 months (after the fall course).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Whitaker, MD, MPH, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Whitaker RC, Herman AN, Dearth-Wesley T, Smith HG, Burnim SB, Myers EL, Saunders AM, Kainz K. Effect of a Trauma-Awareness Course on Teachers' Perceptions of Conflict With Preschool-Aged Children From Low-Income Urban Households: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2019 Apr 5;2(4):e193193. doi: 10.1001/jamanetworkopen.2019.3193. PMID 31026037